CLINICAL TRIAL: NCT04268875
Title: Morphological Parameters of In-stent RESTenosis Assessed and Identified by OCT
Acronym: RESTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Abbott (Industry); Corelab ISIT (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2019 SOUTEYRAND; 2019-A02305-52 (Other: 2019-A02305-52)
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: In-stent Restenosis
Keywords: In-stent restenosis; optical coherence tomography (OCT); coronary angiography
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OCT (Experimental): Patient witch coronary artery disease who has been stented and is hospitalised for stable angina or acute coronary syndrome requiring a further coronary angiogram (regardless of time since implantation or type of the initial stent.
  - Identification of intrastent restenosis during coronary angiography and realisation of an immediate or deferred OCT.
  Interventions: Device: Optical Coherence Tomography (OCT)

INTERVENTIONS:
Device: Optical Coherence Tomography (OCT) — The OCT fibre is an optical fibre catheter containing a lens located at its extremity and positioned distal to the arterial segment to be examined. This is an intracoronary, very high-resolution section technique based on absorption and reflection of close infrared light by stents and tissues.
  OCT analysis is performed during a usual coronary angiography procedure. It is a common technique already used and recommended for intrastent restenosis to establish the mechanism of the process. No new product is being tested. The examination performed is the same.

SUMMARY:
The statistical risk of intrastent stenosis has fallen considerably with the emergence of latest generation coated stents (drug-eluting stents: DES). The number and clinical lifespan of stents implanted over the last twenty-five years, however, explain the fact that restenosis remains a not unusual clinical problem which is expressed as a recurrence of angina or of an acute coronary syndrome (ACS).

The mechanisms involved in this restenosis are multifactorial in nature and differ depending on the type of stent and the time since the restenosis occurred. In symptomatic stent restenosis (angina or acute coronary syndrome), a further angioplasty is usually required, occasionally on an emergency basis. Coronary angiography is often not capable of explaining the mechanical causes of this complication.

Optical coherence tomography (OCT), a high-resolution endocoronary imaging technique can assist in the understanding of the mechanism of restenosis and guide treatment. OCT during angiography provides a detailed analysis of the stents and potential complications: the presence of neoatherosclerosis with or without plaque rupture, intimal hyperplasia, stent under-deployment, stent fracture and distal or proximal progression of the atherosclerosis.

The investigators propose a prospective, multicentre study of all cases of intrastent restenosis, examined by angiography, causing clinical features involving stable angina and acute coronary syndrome. The coronary artery involved will be routinely studied by OCT for a mechanical cause of the intrastent restenosis. The routine use of intrastent OCT may assist in the understanding of causes of restenosis and in the decision on appropriate treatment. There are several possible treatments for restenosis, including balloon angioplasty, coated balloon angioplasty, stenting or aorto-coronary bypass graft surgery.

DETAILED DESCRIPTION:
All stented coronary artery patients hospitalised for stable angina or an ACS requiring a further coronary angiogram (regardless of time since implantation or type of the initial stent) identified to have intrastent restenosis during coronary angiography will be included after being informed and obtaining their informed written consent.

* For cases of stable angina the OCT the will be performed immediately with insertion of the probe distal to the area being studied and then automatic retraction of the fibre during injection of the contrast medium.
* For ACS, the OCT will be performed immediately or on a deferred basis at the discretion of the operator.
* For critical lesions which prevent the OCT fibre passing across the lesion, "soft" predilatation with a 2 mm or smaller balloon is permitted.
* Practical conduct of the OCT:

  * Pullback at baseline state and analysis of the stent with a 5 mm margin proximal and distal to the lesion.
  * OCT analysis: under-deployment of the stent (expansion < 80% of the reference mean surface area), neoatherosclerosis with or without rupture, homogeneous or non-homogeneous hyperplasia, stent fracture and proximal or distal progression of the atherosclerosis.
  * Final pullback in cases of a new angioplasty (balloon angioplasty, angioplasty with a coated balloon or stenting).
* The OCT investigations will be anonymised and registered in their original format with a view to centralised reading (Corelab ISIT, UMR 6284-CNRS, Clermont-Ferrand University).
* The angiography records will be submitted for reading by a panel blinded to the OCT for the purposes of demonstrating the added value of OCT in the fine details of diagnosis and the impact of a treatment decision. The angiograms will be reviewed in a centralised analytical laboratory, which will re-read the procedures blind.
* Patients will be followed up via telephone contact or visit one year after inclusion into the study to record any complications which have developed (possible myocardial infarction, reason, any new revascularisation of the target lesion or another artery and reason for this, any deaths and their causes).

ELIGIBILITY:
Inclusion Criteria:

* Men or women, aged 18 years and over.
* Uncoated, coated or bioresorbable stent restenosis, defined by lumen obstruction of over 50% in the stent and/or within 5 mm proximal or distal to the stent found on coronary angiography.
* Patients treated for an acute coronary syndrome in which restenosis is suspected. It is recommended that OCT be performed after restoring TIMI grade 3 coronary flow in the initial investigation or in a later review at < 7 days.
* Patient informed consent.
* Subscription to a social security system.

Exclusion Criteria:

* Technical inability to perform the OCT (distal lesions, severe chronic renal failure).
* Contraindication to the use of ABBOTT systems when insertion of any type of catheter represents a risk to the patient. The contraindications include the following:

  * Bacteraemia or septicaemia
  * Significant coagulation system abnormalities
  * Patients in whom coronary artery spasm has been diagnosed
  * Patients who do not meet the criteria for coronary artery bypass grafting
  * Patients who do not meet the criteria for percutaneous coronary angioplasty
  * Severe haemodynamic shock or instability
  * Total occlusion
* Life expectancy of under one year for non-cardiac reasons.
* Pregnant or breast-feeding women or women who are fertile and not taking appropriate contraceptives.
* Patients under legal protection or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Characteristics of morphological abnormalities, seen on OCT on millimetre sections of the whole stented segment (5 mm proximally and distally to the stent), potentially responsible for the intrastent restenosis | day 0
  Under-deployment of the stent with percentage under-deployment is defined when the minimum intrastent surface area is less than 80% of the reference surface area.
Characteristics of morphological abnormalities, seen on OCT on millimetre sections of the whole stented segment (5 mm proximally and distally to the stent), potentially responsible for the intrastent restenosis | day 0
  Homogeneous or non-homogeneous intimal hyperplasia.
Characteristics of morphological abnormalities, seen on OCT on millimetre sections of the whole stented segment (5 mm proximally and distally to the stent), potentially responsible for the intrastent restenosis | day 0
  Presence of neoatherosclerosis, with or without rupture.
Characteristics of morphological abnormalities, seen on OCT on millimetre sections of the whole stented segment (5 mm proximally and distally to the stent), potentially responsible for the intrastent restenosis | day 0
  Stent fracture .
Characteristics of morphological abnormalities, seen on OCT on millimetre sections of the whole stented segment (5 mm proximally and distally to the stent), potentially responsible for the intrastent restenosis | day 0
  Progression of the proximal or distal atherosclerosis .

SECONDARY OUTCOMES:
Clinical data | day 0
  time to onset of intrastent restenosis
Clinical data | day 0
  sex
Clinical data | day 0
  age
Clinical data | day 0
  past history of angioplasty
Clinical data | day 0
  myocardial infarction
Clinical data | day 0
  coronary artery bypass grafting
Clinical data | day 0
  multi-vessel disease
Clinical data | day 0
  prosthetic valve
Clinical data | day 0
  heart failure
Clinical data | day 0
  chronic renal failure
Clinical data | day 0
  atrial fibrillation
Clinical data | day 0
  valve disease
Clinical data | day 0
  vascular disease
Clinical data | day 0
  CVA
Clinical data | day 0
  TIA
Cardiovascular risk factors | day 0
  hypertension
Cardiovascular risk factors | day 0
  dyslipidaemia
Cardiovascular risk factors | day 0
  diabetes
Cardiovascular risk factors | day 0
  family history
Cardiovascular risk factors | day 0
  overweight (BMI > 25)
Cardiovascular risk factors | day 0
  smoking habit
Blood sample | day 0, day 365
  Measure of LDL cholesterol
Blood sample | day 0, day 365
  Measure of HDL cholesterol
Blood sample | day 0, day 365
  Measure of triglycerides
Blood sample | day 0, day 365
  Measure of HbA1c
Blood sample | day 0, day 365
  Measure of creatinine
Blood sample | day 0, day 365
  Measure of renal clearance
New revascularisation events | day 365
  new revascularisation event in the target lesion or another artery, myocardial infarctions, deaths and causes of events

CONTACTS AND LOCATIONS:
Overall Officials: Géraud Souteyrand, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (27):
- Université- Hôpital Leuven, Leuven, Belgium
- France (24):
  - CHU Clermont Ferrand, Clermont-Ferrand, Auvergne
  - Clinique la Roseraie, Aubervilliers
  - CH Avignon, Avignon
  - CHRU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHRU Morvan, Brest
  - Hôpital privé saint Martin, Cauro
  - Centre Hospitalier les Hôpitaux de Chartres, Chartres
  - CHRU Grenoble Alpes, Grenoble
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - CHRU Lille, Lille
  - Centre Hospitalier Saint Joseph Saint Luc, Lyon
  - Hospices Civiles Lyon, Lyon
  - AP-HM, Marseille
  - CHRU Nîmes, Nîmes
  - Polyclinique les fleurs, Ollioules
  - AP-HP, Paris
  - Hôpital Privé Institut Mutualiste Montsouris, Paris
  - CHRU Poitiers, Poitiers
  - Clinique Saint Hilaire, Rouen
  - CHRU Strasbourg, Strasbourg
  - Clinique Pasteur Toulouse, Toucy
  - CHRU Toulouse, Toulouse
  - CHRU Hôpitaux de Tours, Tours
- Switzerland (2):
  - CH de Bern, Bern
  - CHUV de Lausanne, Lausanne